CLINICAL TRIAL: NCT06397378
Title: Development and Pilot Testing a Video-based Intervention to Promote HPV Vaccination Among College Students
Brief Title: Engaging College Students in Developing and Testing a Video-based Intervention for HPV Vaccination Promotion
Acronym: HPV videos
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, ChengChing Hiya Liu, Associate Professor, Michigan State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: MSUSTUDY10264; PD66847 (Other: Michigan State University Trifecta Initiative Fubd)
Record Dates: First submitted 2024-04-12; First posted 2024-05-02 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: N/A - Healthy Subjects
Keywords: video intervention; HPV vaccination rate; HPV infection; college students
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Intervention Model Description: This study has been approved by the host university's Biomedical and Health Institutional Review Board (Study ID: STUDY00010264). We propose conducting a two-phase, mixed-methods research project to co-develop a culturally and developmentally appropriate video-intervention (Phase 1) with a Student Advisory Board (SAB) composed of eight college students with diverse background (sex, age, discipline). Once the videos are finalized, we will engage the SAB in the Phase 2 activities aimed to examine the feasibility, acceptability, and preliminary effectiveness of a RCT among college students aged 18-26.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group using CDC factsheet (Active Comparator): We did not develop this intervention. Instead, we will use information from the CDC website on HPV and the HPV vaccine and convert it into a narrated voiceover video to ensure the information is delivered in the same format as our video-based intervention.
  Interventions: Other: CDC HPV Fact Sheet
- Group using videos (Experimental): Ninety-three college students will be randomly assigned to three groups (31 participants in each video group Vs. 30 participants in the CDC group) to watch the created videos. The videos will be presented in randomized order and distributed to participants to minimize bias.
  Interventions: Other: short videos related to HPV and the HPV vaccine

INTERVENTIONS:
Other: short videos related to HPV and the HPV vaccine — Eight college students created and developed four videos on human papillomavirus (HPV) and the HPV vaccine, designed to increase their knowledge and attitude, shape subjective norms, enhance perceived behavioral control, and strengthen intentions to receive the HPV vaccine. Two months after the video intervention, we will follow up with participants to collect their self-reported vaccine uptake status.
  Outcomes will be compared with those of another group whose participants will watch a video presenting CDC information on HPV and the HPV vaccine, adapted into a narrated voiceover format.
  Arms: Group using videos
Other: CDC HPV Fact Sheet — We did not develop this intervention. Instead, we will use information from the CDC website on HPV and the HPV vaccine and convert it into a video with a narrated voiceover format.
  Because our student advisory board will develop four short videos, participants who are randomly assigned to the CDC fact sheet group will watch the converted CDC video four times to ensure that all groups are exposed to the same number of videos.
  Here is the CDC link: https://www.cdc.gov/hpv/vaccines/?CDC_AAref_Val=https://www.cdc.gov/hpv/parents/vaccinesafety.html
  Arms: Group using CDC factsheet

SUMMARY:
HPV vaccines offer hope against HPV-associated cancers for males and females; however, the rate of vaccination has not reached projected public health goals. This study will engage key stakeholders in the research process to co-design and pilot testing a video-based intervention addressing low HPV vaccination rates among college students The intervention and its approach have the potential to reduce health disparities in HPV-associated cancers in young adults via low-cost technology and timely intervention.

DETAILED DESCRIPTION:
Human papillomavirus (HPV) infection is the most common sexually transmitted infection in the United States (U.S.) and a significant public health issue, as almost all sexually active individuals contract it at some point in their lives. Approximately 79 million Americans are infected with HPV, most in their late teens or early 20s. HPV has been found to be associated with cancers for females (e.g., cervical cancer) and males (e.g., penile cancer). The high morbidity, mortality, and economic burden attributed to cancer-causing HPV call for researchers to address this public health concern through vigorous prevention efforts, including HPV vaccination.

HPV-associated cancers could be prevented through vaccination. HPV vaccination is recommended for individuals aged 9-26 years. Economic models have shown that HPV vaccination of adolescents and young adults is cost effective; however, HPV vaccination rates are falling dramatically short of the 80% Healthy People 2030 target recommendation. Young adults such as college students are at higher risk for HPV infection but a significant portion of them is not yet vaccinated against HPV.

Empirical evidence suggests that a lack of awareness and knowledge about HPV and the vaccine, the inconvenience of getting the vaccine, and concern about side effects are main barriers for college students. Current interventions developed to increase HPV vaccination rates are primarily focusing on adolescents as recipients. In the limited interventions developed to address low HPV vaccination rates among college students, most of them only included female college students. In one online RCT study that young adults aged 18-26 were randomized into intervention group (YouTube videos) reported significantly higher vaccination intention compared to comparison group (educational pamphlet); however, the vaccination status was not assessed. College students have advocated for educational videos featuring healthcare providers and peers and sharing videos on YouTube and Instagram.

To our knowledge, this study is the first one of a few video-based interventions co-designed with the main stakeholder-college students to address the low HPV vaccination rates in this at-risk population. This novel intervention is brief, portable, tailored to college students and feasible to fit the intervention into college student's busy schedules.

The investigators will develop a video-based intervention and conduct a pilot randomized trial comparing this intervention to an HPV Fact Sheet developed by CDC. The investigators will target college students aged 18-26 because of their higher risk of contracting HPV infection and low vaccination rates. Aim 1. Develop a developmentally and culturally congruent video-based intervention for college students aged 18-26. The investigators will recruit and form a student advisory board (SAB) consisting of 8-10 college students aged 18-26 to assist with developing four brief HPV education videos (each 2-3 mins long; two will be revised from Co-I's prior research). The advisory board will provide input on the study recruitment plan, assessments, and be involved in data interpretation and dissemination processes. Aim 2. Conduct a pilot randomized controlled trial (RCT) to examine the feasibility (participation rate, retention, intervention fidelity), acceptability (satisfaction) and preliminary efficacy of the intervention to promote HPV vaccination among 80 college students aged 18-26.

Once consented, participants will receive assessments at baseline (T0) using the web-based data collection tool, Qualtrics, before being assigned to one of the two study arms. Participants will be invited to fill out Time 1 (T1) assessment immediately after the intervention (video vs. Fact Sheet) and Time 2 (T2) assessment 2 months after completion of the intervention. The interventions (video and CDC Fact Sheet) and T0-T2 assessments will be administered online. A resource kit including available resources to obtain vaccines will be provided to all participants after T2 assessment. The investigators will also provide the video-based intervention to the students in the comparison arm after T2 assessment should they be interested. Videos will be sent out after participants complete T0. One video will be sent out every 3 days and the intervention (4 videos in total) will be completed in 2-week via emails. Participants in the intervention group can watch the videos at their leisure.

Feasibility will be assessed by response rate (percentage of eligible individuals agreeing to participate), retention (proportion retained through follow-up and complete T0-T2 assessments), intervention fidelity (% of participants watch all stories). Acceptability will be assessed via two Likert-type satisfaction questions. Based on our prior research, the investigators will use the following benchmarks to determine study feasibility as ≥ 80% response rate, ≥ 80% retention rate, ≥ 80% intervention fidelity, and acceptability by a mean satisfaction score ≥ 4.0. Preliminary efficacy will be determined by the % of participants completing the 1st HPV vaccine does within 2 months of completing the intervention.

ELIGIBILITY:
Inclusion Criteria: college students aged 18-26 never receive HPV vaccines able to understand English.

Exclusion Criteria: not able to understand English younger than 18 or older than 26 years old have received HPV vaccines.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Participants' HPV vaccination intention | through study completion, an average of 1 year
  The investigators will assess participants' intention to receive HPV vaccines before and after watching HPV vaccine-related videos, t
Participants' HPV vaccine uptake | through study completion, an average of 1 year
  Participants will be asked if they received any HPV vaccines after watching the videos.
Participants' attitude toward receiving the HPV vaccines | through study completion, an average of 1 year
  Participants' attitude toward receiving HPV vaccines will be assessed before and after watching videos.
Participants' subjective norms | through study completion, an average of 1 year
  Participants' subjective norms regarding receiving HPV vaccines will be assessed before and after watching videos.
Participants' perceived behavioral controls | through study completion, an average of 1 year
  Participants' perceived behavioral control regarding receiving HPV vaccines will be assessed before and after watching videos.
Participants' satisfaction | through study completion, an average of 1 year
  participants' satisfaction about the interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan State University, East Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD including individuals' intention to receive the HPV vaccines and developed videos can be shared upon request.
Supporting Information: Study Protocol
Time Frame: December 2025
Access Criteria: To increase the robustness of the study design and results, the team member who handles data and analysis will be blinded to the assignment of participants in the respective study arms. Each participant will be assigned a unique ID linked to respective random group assignments. One unblinded team member will be selected to make reminder calls; this staff member will not be involved in intervention delivery or data entry, cleaning, or analysis. The PI will closely monitor the procedures to ensure high treatment fidelity.
URL: https://nursing.msu.edu

REFERENCES:
- [Derived] Liu C, Chen AC, Rhodes N, Ewoldsen D, Arcoleo K. Evaluating the preliminary effectiveness of a video-based intervention for HPV vaccination promotion among college students aged 18-26: study protocol for a pilot randomised controlled trial. BMJ Open. 2025 Nov 16;15(11):e102235. doi: 10.1136/bmjopen-2025-102235. PMID 41248380